CLINICAL TRIAL: NCT03567850
Title: Problem Solving Skills Training in Adult Cancer Survivors: Bright IDEAS-AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 65518
Record Dates: First submitted 2018-05-31; First posted 2018-06-26 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants assigned to the intervention arm will receive Problem Solving Skills Training (PSST) consisting of eight one-hour individual weekly sessions.
  Interventions: Behavioral: Problem solving Skills Training
- Control Arm (Active Comparator): Care As Usual Group (CAU): Participants randomized to the CAU group will be observed under naturalistic conditions. Both PSST and CAU participants and their clinicians (PCP and oncology providers) will be allowed to use any clinically appropriate medical and behavioral care without restriction (e.g., care management, rehabilitation, behavioral therapy, palliative care) or refer patients to social and community services (e.g., peer support, county cancer services program or aging services). The CAU participants will undergo the same evaluation protocol as the PSST group
  Interventions: Behavioral: Problem solving Skills Training

INTERVENTIONS:
Behavioral: Problem solving Skills Training — Participants will be encouraged to identify specific problems particularly relevant to them and to their family's situation (instead of providing them with standardized examples) to be discussed and "solved" during the PSST sessions. The eight sessions of PSST will be organized in a systematized, therapeutic manner. Session 1 will be face-to-face and devoted to rapport building and understanding relevant social and medical information. The therapist (RA) will introduce PSST and the Bright IDEAS paradigm, present worksheets to guide PSST homework assignments, and give an overview of subsequent sessions. Starting at session 2, participants will continue training over the phone, with the same general structure and format. In sessions 2-7, the therapist and patient, with a supportive other (SO) if available, will review the patient's identified problems and work on application of problem-solving strategies and skills learned earlier.

SUMMARY:
The aim of this 2-year study will assess the acceptability and feasibility of offering Problem Solving Skills Therapy (PSST) to cancer survivors and their caregivers focusing on the highest risk patients with distress.

DETAILED DESCRIPTION:
At Roswell Park Comprehensive Cancer Center, in collaboration with the University at Buffalo School of Public Health and Health Professions and the University of Rochester, we are looking for adult cancer patients to participate in our new project designed to facilitate recovery from cancer and help cancer survivors lead better, more productive lives. The ideal subjects are individuals who have completed treatment for stage I-III cancer and speak English. Participants will be randomized into two groups: 8 weekly 1-hour long sessions of problem solving skills therapy delivered by a trained therapist vs. care as usual. Bright IDEAS Adult Cancer (Bright IDEAS-AC) therapy will be delivered in the most patient-friendly way. Sessions will be face-to-face at the location of patient choice (hospital, clinic, or participant's home) or over the phone. A supportive other or caregiver is also invited to participate in this study. This project does not involve any experimental drugs and does not affect the regular care or patient relationship with doctor(s).

At the time of enrollment, after 3 months and after 6 months, all participants in the intervention and control arms, as well as any participating supportive others/caregivers will be asked about their healthcare utilization since the last assessment including primary care, specialist and emergency department visits and any hospital stays. During the same three time points, both patients and supportive others/caregivers will be asked to fill in 4 short questionnaires assessing their problem solving skills, health status, mood and function

ELIGIBILITY:
Inclusion Criteria:

* stage I-III Colorectal Cancer, Breast, Bladder or Prostate Cancer
* meet the screening criteria for psychological distress (NCCN Distress >2)
* be able to speak English
* have a 5-year survival rate of 50% or greater as deemed by their oncologist, surgeon,or other relevant attending physician (suggesting a reasonable rate of cure or prolonged medical survival with state-of-the-art medical care)
* be willing to provide written informed consent to participate in the study which includes several clinical evaluations, provide access to medical records/PCP, and allow all interviews and PSST therapy sessions to be audiotaped.
* Among patients treated in the urban centers, we will specifically target patients who live more than 40 miles away from the clinic as they are more likely to experience problems with access to care.
* Age 21 or older

Exclusion Criteria:

* a diagnosis of mental retardation,
* and/or acute suicidal behavior

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekaternia Noyes, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Noyes K, Zapf AL, Depner RM, Flores T, Huston A, Rashid HH, McNeal D, Constine LS, Fleming FJ, Wilding GE, Sahler OJZ. Problem-solving skills training in adult cancer survivors: Bright IDEAS-AC pilot study. Cancer Treat Res Commun. 2022;31:100552. doi: 10.1016/j.ctarc.2022.100552. Epub 2022 Mar 25. PMID 35358820

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: Care As Usual Group (CAU): Participants randomized to the CAU group will be observed under naturalistic conditions.
  Problem solving Skills Training: Participants will be encouraged to identify specific problems particularly relevant to them and to their family's situation (instead of providing them with standardized examples) to be discussed and "solved" during the PSST sessions. The eight sessions of PSST will be organized in a systematized, therapeutic manner. Session 1 will be face-to-face and devoted to rapport building and understanding relevant social and medical information. The therapist (RA) will introduce PSST and the Bright IDEAS paradigm, present worksheets to guide PSST homework assignments, and give an overview of subsequent sessions. Starting at session 2, participants will continue training over the phone, with the same general structure and format. In sessions 2-7, the therapist and patient, with a supportive other (SO) if available, will review the patient's identified problems and work on application of problem-solving strategies and skills learned earlier.
Period: Overall Study
Arm/Group | Intervention | Control Arm
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control Arm | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.4) | 62.3 (8.4) | 63.1 (8.9)
Age, Customized [Count of Participants; unit: Participants]
  Age: 40-49 | 2 | 2 | 4
  Age: 50-59 | 6 | 6 | 12
  Age: 60-69 | 13 | 12 | 25
  Age: 70-79 | 2 | 4 | 6
  Age: 80+ | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 22 | 22 | 44
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Marital Status [Count of Participants; unit: Participants]
  Single | 2 | 0 | 2
  Married | 15 | 18 | 33
  Divorced | 7 | 6 | 13
  Other | 1 | 1 | 2
Diagnosis [Count of Participants; unit: Participants]
  Colon and Rectal Cancer | 10 | 10 | 20
  Breast Cancer | 10 | 11 | 21
  Prostate Cancer | 5 | 4 | 9
Is Caregiver Also Participating [Count of Participants; unit: Participants]
  No | 20 | 13 | 33
  Yes | 5 | 12 | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Physical Health of Patient at Enrollment
Description: From all patients in the intervention and control arms, we will collect patient on physical health using the Functional Assessment of Cancer Therapy - disease specific.
  FACT-G is a 27-item questionnaire designed to measure four domains of health-related quality of life in cancer patients based on the past 7 days: physical, social, emotional, and functional well-being (score range is 1-108; higher scores indicate better quality of life). The scale's ability to discriminate patients on the basis of performance status and hospitalization status supports its sensitivity. It has also demonstrated sensitivity to change over time. Differences of 5-7 points are considered clinically significant.
Time Frame: At enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 25 | 22
score on a scale | 77.2 (21.3) | 82.7 (16.7)

2. Primary Outcome: Behavioral Health of Patient
Description: From all patients in the intervention and control arms, we will collect patient self-report data on problem solving skills,using the Social Problem-Solving Inventory-Revised (SPSI-R)
  SPSI-R is a 25-item self-report tool linked to a multidimensional model of problem-solving skills. SPSI-R:S has been demonstrated to have strong reliability and validity estimates. The scale includes 5 sub-scales grouped into two decision-making styles: constructive (Positive Problem Orientation and Rational Problem Solving) and dysfunctional (Negative Problem Orientation, Impulsivity/ Carelessness, and Avoidance). Each subscale and the total SPSI-R:S scores are expressed on a 0-20 scale; higher scores indicate better skills.
Time Frame: At time of enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 25 | 25
score on a scale | 12.2 (3.7) | 11.7 (3.7)

3. Primary Outcome: Mean Change in Physical Health From Baseline to 3-months
Description: From all patients in the intervention and control arms, we will collect patient on physical health using the Functional Assessment of Cancer Therapy - Disease Specific (FACT)
  FACT-G is a 27-item questionnaire designed to measure four domains of health-related quality of life in cancer patients based on the past 7 days: physical, social, emotional, and functional well-being (score range is 1-108; higher scores indicate better quality of life). The scale's ability to discriminate patients on the basis of performance status and hospitalization status supports its sensitivity. It has also demonstrated sensitivity to change over time. Differences of 5-7 points are considered clinically significant.
  The mean change was calculated as the difference between the 3-month measurement and the baseline measurement.
Time Frame: At 3 months
Population: A total of 3 patients did not fully complete the FACT-G survey at 3-months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 25 | 25
score on a scale
  baseline | 77.2 (21.3) | 82.7 (16.7)
  3-months: number analyzed (Participants) | 22 | 25
  3-months | 82.4 (19.6) | 82.4 (20.2)

4. Primary Outcome: Mean Change Physical Health of Patient at 12 Months
Description: From all patients in the intervention and control arms, we will collect patient on physical health using the Functional Assessment of Cancer Therapy (FACT)
  FACT-G is a 27-item questionnaire designed to measure four domains of health-related quality of life in cancer patients based on the past 7 days: physical, social, emotional, and functional well-being (score range is 1-108; higher scores indicate better quality of life). The scale's ability to discriminate patients on the basis of performance status and hospitalization status supports its sensitivity. It has also demonstrated sensitivity to change over time. Differences of 5-7 points are considered clinically significant.
Time Frame: At 12 months
Population: A total of 6 patients did not complete the 12-month FACT-G survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 25 | 25
score on a scale
  baseline | 77.2 (21.3) | 82.7 (16.7)
  12-months: number analyzed (Participants) | 20 | 24
  12-months | 87.1 (21.5) | 82.3 (18.9)

5. Primary Outcome: Mean Change in Behavioral Health of Patient at 3 Months
Description: as for outcome 2
Time Frame: At 3 months
Population: A total of 3 patients did not complete the SPSI-R at 3-months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 25 | 25
score on a scale
  baseline | 12.2 (3.7) | 11.7 (3.7)
  3-months: number analyzed (Participants) | 22 | 25
  3-months | 13.4 (3.8) | 11.6 (4.2)

6. Primary Outcome: Mean Change in Behavioral Health of Patient at 12 Months
Description: as for outcome 2
Time Frame: At 12 months
Population: A total of 6 subjects did not complete the SPSI-R at 12-months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 25 | 25
score on a scale
  baseline | 12.2 (3.7) | 11.7 (3.7)
  12-months: number analyzed (Participants) | 20 | 24
  12-months | 13.8 (3.1) | 11.7 (4.5)

7. Primary Outcome: Healthcare Utilization of Patients
Description: From all patients in the intervention and control arms, we will collect patient self-report data by asking the patients about their healthcare utilization since the last study assessment including primary care, specialist and ED visits, use of supportive services and any hospital stays.
Time Frame: At 12 months
Population: 6 patients did not complete these questions on the final follow-up survey.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 20 | 24
visits
  Number of Hospital Visits | 0.0 (0.0) | 0.4 (0.9)
  Number of Emergency Room Visits | 0.0 (0.0) | 0.3 (0.9)
  Number of Ambulatory Services Used | 6.5 (4.7) | 5.7 (3.9)

ADVERSE EVENTS:
Time Frame: Subjects were followed for 12 months after randomization.
Arm/Group | Intervention | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT03567850/Prot_SAP_000.pdf